CLINICAL TRIAL: NCT04906044
Title: Total Neoadjuvant Treatment Plus PD-1 in Mid-Low Locally Advanced Rectal Cancer (STARS-RC03)
Brief Title: Total Neoadjuvant Treatment Plus PD-1 in Mid-Low Locally Advanced Rectal Cancer
Acronym: STARS-RC03
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS-RC03
Record Dates: First submitted 2021-05-10; First posted 2021-05-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tislelizumab; Locally Advanced Rectal Cancer; Total Neoadjuvant Treatment; PD-1
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Neoadjuvant Treatment combined with Sintilimab (Experimental)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab combined withTotal Neoadjuvant Treatment

SUMMARY:
There have been many high-quality research publications, including the TNT model of short-term radiotherapy combined with consolidation chemotherapy, and the TNT model of three-drug combination with neoadjuvant chemotherapy with higher treatment intensity combined with CRT. All have achieved better tumor regression and tumor regression than the standard CRT model. The higher pCR rate reduces the recurrence and metastasis events, improves the prognosis, and strives for more opportunities for organ function preservation. Can the TNT model combined with immunotherapy further increase the cCR rate? Whether immunotherapy can bring further survival benefits to patients who develop CR after neoadjuvant therapy (especially W&W after cCR), it is also necessary to carry out corresponding clinical research. We designed this study for patients with mid-to-low and locally advanced rectal cancer who want to be able to preserve the anus. TNT mode combined with PD-1 immunotherapy is given before surgery, and TME surgery is performed on patients who have not reached cCR or who still require surgery. It provides sufficient evidence for the safety and effectiveness of preoperative neoadjuvant therapy for PD-1 in low- and middle-level locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients and their families are able to understand and are willing to participate in this clinical study, and sign an informed consent form.
2. Age: 18~80 years old, no gender limit;
3. Pathologically diagnosed rectal adenocarcinoma: differentiated into Grade 1-3, that is, high, medium, and poorly differentiated tubular adenocarcinoma;
4. The initial MRI partial phases are: 1) Local intermediate risk: T3c/d or N1-2 (carcinoma nodules) or very low position or EMVI+ or MRF 1-2mm, without external iliac, total iliac, obturator, main abdomen Arterial lymph node metastasis; 2) Local high risk: T4 or MRF+ or lateral lymph node positive.
5. The distance from the lower edge of the tumor is below the reflex of the peritoneum (MRI evaluation);
6. No distant transfer;
7. ECOG PS score 0-1 within 7 days before the first medication;
8. Hepatitis B Surface Antigen (HBsAg) (-) and Hepatitis B Core Antibody (HBcAb) (-). If HBsAg (+) or HBcAb (+), hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be less than 1000 copies/mL or 200 IU/mL before entering the group.
9. HCV antibody (-)
10. The main organ function is normal.
11. No history of pelvic radiotherapy;
12. No history of rectal cancer surgery or chemotherapy;
13. Not accompanied by systemic infections requiring antibiotic treatment;
14. Heart, lung, liver, and kidney functions can tolerate surgery;
15. Others, based on the results of previous medical history, vital signs, physical examination or laboratory examination, the research doctor judges that you are suitable for participating in this clinical study.

Exclusion Criteria:

1. Recurrent rectal cancer;
2. The patient cannot tolerate enhanced nuclear magnetic examination;
3. Patients who are planning to undergo or have previously received organ or bone marrow transplantation;
4. Myocardial infarction or poorly controlled arrhythmia (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females) occurred within 6 months before the first medication (QTc interval is calculated by Fridericia formula);
5. Existence of NYHA standard grade III to IV cardiac insufficiency or color Doppler ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
6. Human immunodeficiency virus (HIV) infection;
7. Suffer from active tuberculosis;
8. Past and present patients with interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc., which may interfere with the detection and treatment of suspected drug-related lung toxicity;
9. There is a known active or suspicious autoimmune disease. Except those who were in a stable state of the disease at the time of enrollment (no need for systemic immunosuppressive therapy);
10. Received treatment with live vaccines within 28 days before the first administration; except for inactivated viral vaccines for seasonal influenza;
11. Patients who need to receive systemic corticosteroids (> 10 mg/day curative dose of prednisone) or other immunosuppressive drugs within 14 days before the first medication or during the study period. However, the following conditions are allowed to enter the group: in the absence of active autoimmune diseases, patients are allowed to use topical or inhaled steroids, or adrenal hormone replacement therapy with a dose ≤ 10 mg/day prednisone curative dose;
12. Any active infection that requires systemic anti-infective treatment occurs within 14 days before the first administration; except for receiving preventive antibiotic treatment (such as preventing urinary tract infection or chronic obstructive pulmonary disease);
13. Have received other antibody/drug treatments against immune checkpoints in the past, such as PD-1, PD-L1, CTLA4, etc.;
14. Known to have a history of severe allergies to any monoclonal antibody or research drug excipients;
15. In the past 5 years, patients have suffered from malignant tumors whose survival rate is significantly lower than the historical data of our rectal cancer survival rate (properly treated basal cell carcinoma, skin squamous cell carcinoma, small kidney cancer, breast cancer, and papillary thyroid carcinoma are not included here. range);
16. The patient has had arterial embolism diseases in the past 6 months, such as angina pectoris, MI, TIA, CVA, etc.;
17. Have received other types of anti-tumor or experimental treatments;
18. The patient is a female during pregnancy or lactation;
19. The patient has other diseases or abnormal mental states, which may affect the patient's participation in this study;
20. There are patients who may increase the risk of participating in research and research medication, or other severe, acute and chronic diseases, who are not suitable for clinical research based on the judgment of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of serious adverse events | 1 year
  Any treatment-related grade 3 or higher non-hematological adverse event determined by CTCAE version v 4.03.

SECONDARY OUTCOMES:
Complete response rate (CR) | one week after Last medication
  defined as cCR or pCR achieved after neoadjuvant therapy.
Neoadjuvant colorectal cancer (NAR) score | One week after the surgery
  NAR score is a continuous scale with 24 possible discrete scores, ranging from 0 to 100. In this patient cohort, low scores were defined as <8, median values were 8-16, and high scores were> 16, and the corresponding 5-year OS was 92%, 89%, and 68%, respectively. A higher score is associated with a worse prognosis.
Tumor downgrading rate | One week after surgery
  the rate of downgrading confirmed by MRI
3-year non-local regeneration disease-free survival (NR-DFS) | 3 years from the date of receiving neoadjuvant therapy
  It is defined as the time of death, local recurrence after radical resection, and any form of distant metastasis within 3 years from the date of receiving neoadjuvant therapy. The local regeneration of the tumor that can be rescued after non-surgical treatment is not regarded as a local recurrence, nor is it counted as a positive event.
3 years disease-free survival | 3 years from the date of receiving neoadjuvant therapy
  3 years disease-free survival
5 years disease-free survival | 5 years from the date of receiving neoadjuvant therapy
  5 years disease-free survival
3-year local recurrence rate | 3 years from the date of receiving neoadjuvant therapy
  3-year local recurrence rate
3 years overall survival | 3 years from the date of receiving neoadjuvant therapy
  3 years overall survival
5 years overall survival | 5 years from the date of receiving neoadjuvant therapy
  5 years overall survival
QLQ-C30 score | up to 12 months
  QLQ-C30（Quality of Life Questionnaire C30）
QLQ-C29 | up to 12 months
  QLQ-C29(Quality of Life Questionnaire C29）
Low Anterior Resection Syndrome | up to 12 months
  LARS score（Low Anterior Resection Syndrome Questionnaire）
IPSS score | up to 12 months
  IPSS score（International Prostate Symptom Score）
CIPE score | up to 12 months
  CIPE （Chinese Index of sexual Function for premature Evaluation,CIPE）score
Quality of life and function assessment | up to 12 months
  IIEF-5(international questionnaire of erectile function-5)score
FEFSI-6 score | up to 12 months
  FEFSI-6 score
Wexner score | up to 12 months
  Wexner incontinence score

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No